CLINICAL TRIAL: NCT02953574
Title: Daily Sleep Enhancement for Hospitalized People With Dementia Following a 7 Step Nursing Protocol: a Quasi-experimental Pilot Study
Brief Title: Daily Sleep Enhancement for Hospitalized People With Dementia Following a Nursing Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-00780
Record Dates: First submitted 2016-10-20; First posted 2016-11-03 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Sleep; Dementia
Keywords: geriatric nursing
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- daily sleep enhancement nursing protocol (Experimental): A 7 step nursing protocol. Each step is daily provided to the demented patient through a nurse by bedtime.
  Step 1: serve a late snack Step 2: evening care (brush teeth, get pyjama on, go to toilette) Step 3: note and treat physical circumstances that restrain sleep (pain, obstipation,...) Step 4: ensure comfortable position abed Step 5: assist to eliminate stressful situation (calm, reorientating conversation) Step 6: turn off the light Step 7: care for a silent environment (turn off Television, radio and "do not disturb"-sign at the door)
  Interventions: Procedure: daily sleep enhancement nursing protocol
- usual nursing care (No Intervention)

INTERVENTIONS:
Procedure: daily sleep enhancement nursing protocol
  Arms: daily sleep enhancement nursing protocol

SUMMARY:
The purpose of this study is to determine if the daily performance of a 7 step bedtime nursing protocol for hospitalized people living with dementia is feasible and if it has an effect on bedtime and daytime variables.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dementia of any severity and type
* Allocation to geriatric rehabilitation treatment

Exclusion Criteria:

* sleep related respiratory or moving related disorders or Parasomnia
* delirium
* end of life care

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Bedtime in minutes | Daily for up to 14 days from date of giving informed consent to hospital discharge
  Protocol of daily bedtime

SECONDARY OUTCOMES:
Sleeps through the night consistently, 5 point ordinal scale from "severe compromised" to "not compromised" | Every second day for up to 14 days from date of giving informed consent to hospital discharge
  Subitem of the Outcome 'Sleep' from the Nursing Outcome Classification (NOC)
  Scale:
  1. severe compromised
  2. substantial compromised
  3. moderate compromised
  4. mild compromised
  5. not compromised
Inappropriate napping, 5 point ordinal scale ranging from "sever" to "none" | Every second day for up to 14 days from date of giving informed consent to hospital discharge
  Subitem of the Outcome 'Sleep' from the Nursing Outcome Classification (NOC)
  Scale:
  1. severe
  2. substantial
  3. moderate
  4. mild
  5. none
Cognitive performance (Mini-mental-status-test score) | Once in first three days after giving informed consent and another time 7 or 14 days later
  Mini-mental-status-test score (range 0-30). Any score greater than or equal to 24 points (out of 30) indicates a normal cognition.
  Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment
Physical performance measured with the Handgrip strength test | Once in first three days after giving informed consent and another time 7 or 14 days later
  Handgrip strength in Pascal
Use of drugs promoting sleep (sedative neuroleptics, hypnotics, sedative antidepressant in the time between 18:00-24:00) (nominal variable: yes or no) | day 1,2 and day 6,7 or 13,14
  Medical charts review for sedative neuroleptics (e.g. Quetiapine, Haloperidol), sedative antidepressives (e.g. Trazodon), hypnotics present (Benzodiazepines, benzodiazepine-like drugs) in the time between 18:00-24:00 (nominal variable: yes or no )
Medical chart review for discharge domicile after hospitalisation (nursing home, home, other institution, other) | day 7 or 14
  Domicile after hospital discharge

OTHER OUTCOMES:
Application frequency of the nursing (ritual) protocol | Every day for up to 14 days from date of giving informed consent to hospital discharge
  Daily protocol of the received and of the refused interventions of the nursing ritual (frequency)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Burkhalter, Dr. sc. med., Principal Investigator — Center of Sleep Medicine

IPD SHARING:
Plan to Share IPD: No